CLINICAL TRIAL: NCT02364011
Title: Clinical and Biomechanical Outcomes Following Total Knee Arthroplasty
Brief Title: Outcomes Following Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Pelt, Principle Investigator, University of Utah
Other Study IDs: 75446
Record Dates: First submitted 2015-02-09; First posted 2015-02-16 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis
Keywords: Biomechanics; Primary Total Knee Arthroplasty; TKA Bearings; Osteoarthritis; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this investigation is to determine both patient-reported and performance-based outcomes, specifically muscle function and kinematic/kinetic outcomes, between four different surgical total knee prostheses in individuals following TKA. Change scores will be determined based on patient-reported outcomes, kinematic/kinetic data, knee extension strength/power, static/dynamic balance control, mobility measures and functional performance testing during functional tasks (i.e. walking, ascending/descending stairs, sit-to-stand). After evaluating the pattern of change in lower-extremity function, the investigators will be better prepared to address residual functional impairments and prognostic factors linked to maximal recovery over two years.

ELIGIBILITY:
Inclusion Criteria:

* adults > 40 years of age that are scheduled for primary TKA
* if they have had a previous TKA, it needs to have been performed on the opposite leg at least 3 months prior to the current TKA
* willing to return for follow-up visits and should be willing and able to be transported from the UOC to the Skeletal Muscle Exercise Research Facility (SMERF), in the Department of Physical Therapy study site for scheduled research follow-up appointments

Exclusion Criteria:

* adult with previous additional orthopaedic, neurological, visual or surgical conditions that may affect gait or balance

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the University of Utah for TKA surgical procedure
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-11; Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcome Scores following TKA | Follow Up Visits up to 2-Years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Pelt, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States